CLINICAL TRIAL: NCT00792064
Title: Systematic Evaluation of Predictors of Quality of Life in the Long-term After Solid Organ Transplantation- a Prospective Cohort Study
Brief Title: Systematic Evaluation of Predictors of Quality of Life in the Long-term After Solid Organ Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Dr. rer. biol. hum. Christiane Kugler, Hannover Medical School
Other Study IDs: IRB No_378
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Organ Transplantation; Anxiety; Depression
Keywords: quality of life; adverse effects
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Kidney-Tx-recipients
- 2: Liver-Tx-recipients
- 3: Heart-Tx-recipients
- 4: Lung-Tx-recipients

SUMMARY:
A systematic evaluation of predictors of health related quality of life (HRQoL) leads to multiple level of data analysis. The aim of the herein described observational project is to create a transplant patients registry on psychosocial outcomes and to evaluate longitudinally predictors of HRQoL after different types of solid organ transplantation in the long-term. A sample size of 700 participants consisting of all solid organ types is envisioned. Data will be compared with published healthy normative data. Data Evaluation of predictors of HRQoL may guide development of tailored interventions to reduce complications and to further improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up at our outpatient clinics
* Written informed consent
* Sufficient German language skills to read and answer a battery of questionnaires
* Min 18 years

Exclusion Criteria:

* Illiteracy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients immediately after solid organ transplantation
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2009-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
HRQoL after transplantation | 5 yrs

SECONDARY OUTCOMES:
Social re-integration | 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Kugler, PhD, Principal Investigator — Clinic for Cardiac, Thoracic, Transplantation and
Locations (1):
- Hannover Medical School, Clinic für cardias, thoracic, transplantation and vascular surgery, Hanover, Germany